CLINICAL TRIAL: NCT05160922
Title: CRIZOTINIB MASTER PROTOCOL: AN OPEN-LABEL CONTINUATION STUDY FOR PARTICIPANTS CONTINUING FROM PFIZER-SPONSORED CRIZOTINIB CLINICAL STUDIES
Brief Title: Crizotinib Continuation Clinical Study
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A8081075; 2024-511128-15-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-12-06; First posted 2021-12-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: NSCLC; ALCL; IMT
Keywords: crizotinib; Xalkori; Anaplastic Lymphoma Kinase; ALK; ROS1; NSCLC; Non-small Cell Lung Cancer; ALCL; anaplastic large cell lymphoma; IMT; inflammatory myofibroblastic tumour
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lymphoma, Large-Cell, Anaplastic; Granuloma, Plasma Cell | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- crizotinib (Other): crizotinib oral treatment
  Interventions: Drug: crizotinib

INTERVENTIONS:
Drug: crizotinib — crizotinib oral treatment
  Other Names: XALKORI

SUMMARY:
The purpose of this continuation study is to provide continued access to crizotinib treatment for eligible participants from a current Pfizer sponsored crizotinib clinical study that is planned to close.

DETAILED DESCRIPTION:
Participants not previously enrolled or who have discontinued study treatment or safety follow-up in a current Pfizer sponsored crizotinib clinical study are not eligible for participation in this continuation study.

ELIGIBILITY:
Participants must meet the following key inclusion criteria to be eligible for enrollment into the study:

1. Any participant who is receiving crizotinib and deriving clinical benefit (as determined by their doctor) in a Crizotinib Study which is planned to close.
2. Participants must agree to follow the reproductive criteria as outlined in protocol.
3. No ongoing Grade ≥3 or intolerable Grade 2 AEs considered to be related to crizotinib treatment, except for those laboratory eligibility criteria described in Inclusion #4.
4. Adult Participants (≥18 years): Adequate hepatic and bone marrow function. Stable renal function for at least 14 days.

Pediatric Participants (<18 years): Adequate hepatic and bone marrow function. Stable renal function for at least 14 days.

Exclusion Criteria

Participants with any of the following characteristics/conditions will be excluded:

1. Female participants who are pregnant or breastfeeding.
2. Any medical reason that, in the opinion of the investigator or sponsor, precludes the participant from inclusion in the study.

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2028-03-21 (Estimated); Study Completion 2028-03-21 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events leading to permanent discontinuation of study intervention | Baseline up to approximately 5 years
  Safety data collection in this study will permit further characterization of the safety profile of crizotinib.
Number of serious adverse events reported for all participants | Baseline up to approximately 5 years
  Safety data collection in this study will permit further characterization of the safety profile of crizotinib.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- China (9):
  - Cancer Hospital Chinese Academy of Medical Science, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Province Oncology Hospital, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer center, Guangzhou, Guangdong
  - Jilin Cancer Hospital, Changchun, Jilin
  - West China Hospital of Sichuan University, Wuhou District, Sichuan
  - The First Affiliated Hospital of College of Medicine,Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Guangzhou Medical University., Guangzhou
  - Shanghai Chest Hospital, Shanghai
- ASST Monza, Monza, MB, Italy
- National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken, Japan
- Limited Liability Company "EuroCityClinic", Saint Petersburg, Russia
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A8081075